CLINICAL TRIAL: NCT06990997
Title: Effects of Aphasia Identification Cards on Comprehension of Aphasic Language by Unfamiliar Communication Partners
Brief Title: Effects of Aphasia Identification Cards on Service Workers' Comprehension of People With Aphasia
Acronym: PAUSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Amherst (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Jennifer Mack, Assistant Professor, University of Massachusetts, Amherst
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB #5783; 1R21DC021233-01A1 (NIH)
Record Dates: First submitted 2025-05-01; First posted 2025-05-25 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Aphasia
Keywords: Aphasia; Communication partner; Service worker; Language processing; Language comprehension; aphasia identification card; eye-tracking
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aphasia Identification Card (Experimental): Participants will view an aphasia ID card for a speaker with aphasia. The card will disclose the speaker's aphasia, define aphasia, and request time to communicate.
  Interventions: Behavioral: Aphasia identification (ID) card
- No Card (No Intervention): Participants in this arm will not receive an intervention.

INTERVENTIONS:
Behavioral: Aphasia identification (ID) card — Participants will view an aphasia ID card for a speaker with aphasia. The card will disclose the speaker's aphasia, define aphasia, and request time to communicate.
  Arms: Aphasia Identification Card

SUMMARY:
The goal of this clinical trial is to learn whether healthy volunteers are more successful at understanding people with aphasia if they have first viewed an aphasia identification (ID) card. The main questions this study aims to answer are:

* Does viewing an aphasia ID card improve healthy volunteers' understanding of the language errors made by people with aphasia?
* Does viewing an aphasia ID card improve healthy volunteers' understanding of people with aphasia who make long pauses in their speech?

Researchers will compare aphasia ID cards to a control condition (no ID card) to see whether aphasia ID cards improve healthy volunteers' understanding.

Healthy volunteers will visit the study site for a single session (about 2 hours long). During the session they will:

* Complete brief tests of their vision, hearing and thinking
* Listen to sentences produced by a speaker with aphasia while their eye movements are recorded
* Complete a survey about the experience of listening to the speaker with aphasia

DETAILED DESCRIPTION:
People with aphasia often experience challenges conveying their thoughts to unfamiliar communication partners, which is critical for living independently and building new social connections. This line of research has two long-term objectives: to improve unfamiliar communication partners' comprehension of people with aphasia, and to support people with aphasia in advocating for their communication needs. This project addresses these goals with a focus on service workers, who interact directly with customers to provide goods, services, or information. Being understood by service workers is often necessary to complete essential tasks such as purchasing food and picking up medication. This project investigates whether service workers comprehend speakers with aphasia more accurately when they have first read an aphasia identification (ID) card. Aphasia ID cards contain written self-advocacy statements that disclose the speaker's aphasia, define aphasia, and provide guidance on how to communicate successfully. These statements have been shown to improve unfamiliar communication partners' attitudes (knowledge about aphasia, emotions, and behavior), which improves communication experiences for people with aphasia. This project tests the central hypothesis that, by improving unfamiliar communication partners' attitudes, aphasia ID cards facilitate key language processes that improve their comprehension of people with aphasia. This randomized controlled trial will enroll 160 service workers. Half of the service workers will view an aphasia ID card for a speaker with aphasia, and half will not. Then, all service workers will complete tasks measuring their attitudes, language processing, and comprehension of service requests (i.e., requests for goods, services, or information) produced by speakers with aphasia. Eye-tracking will be used to measure key language processes that take place while service workers listen to the service requests. The Specific Aims are to investigate how viewing an aphasia ID card affects service workers' attitudes, language processing, and comprehension when people with aphasia produce long pauses (Aim 1) and paraphasias (word-retrieval errors) (Aim 2). By rigorously investigating the effects of aphasia ID cards on service workers' attitudes, language processing, and comprehension, this project will contribute to the long-term goals of improving unfamiliar communication partners' comprehension and helping people with aphasia self-advocate effectively.

ELIGIBILITY:
Inclusion Criteria:

* Adult age 18-59
* Currently employed as a service worker
* Understand spoken and written English well
* High school diploma or equivalency
* Normal vision or corrected vision with glasses or contact lenses

Exclusion Criteria:

* Language disorder
* Hearing impairment
* Intellectual disability
* History of acquired neurological disorder (e.g., stroke or moderate/severe brain injury)

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-09-22 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Comprehension accuracy for sentences with long pauses in the Service Request Comprehension Task | 5 minutes post-intervention
  Percent correct mouse-click responses on the Service Request Comprehension Task for sentences with long pauses. The Service Request Comprehension Task measures participants' comprehension and processing of language produced by a speaker with aphasia.
Comprehension accuracy for sentences with paraphasias in the Service Request Comprehension Task | 5 minutes post-intervention
  Percent correct mouse-click responses on the Service Request Comprehension Task for sentences with paraphasias (word-retrieval errors). The Service Request Comprehension Task measures participants' comprehension and processing of language produced by a speaker with aphasia.

SECONDARY OUTCOMES:
Visual attention during long pauses in the Service Request Comprehension Task | 5 minutes post-intervention
  Mean proportion of time in which the participant gazes at task-relevant pictures during long pauses, indicating attention to task. The Service Request Comprehension Task measures participants' comprehension and processing of language produced by a speaker with aphasia.
Linguistic integration of words immediately following long pauses in the Service Request Comprehension Task | 5 minutes post-intervention
  Mean proportion of time in which the participant gazes at the target picture during words immediately following long pauses, indicating linguistic integration of those words. The Service Request Comprehension Task measures participants' comprehension and processing of language produced by a speaker with aphasia.
Implicit repair of paraphasias in the Service Request Comprehension Task | 5 minutes post-intervention
  Mean proportion of time in which the participant gazes at the target picture in the 1000 ms following paraphasias (word-retrieval errors), indicating implicit repair of the speaker's errors. The Service Request Comprehension Task measures participants' comprehension and processing of language produced by a speaker with aphasia.
Rating of own patience on the Attitude Survey | 0 minutes (immediately) post-intervention, 45 minutes post-intervention
  Rating scale, 0-100 scale with question "When listening to the speaker, I felt _____", with endpoints of "impatient" on the zero side and "patient" on the 100 side. Higher scores mean a better outcome. The Attitude Survey measures participants' knowledge, beliefs, and emotions relating to listening to a speaker with aphasia.
Rating of speaker with aphasia's intelligence on the Attitude Survey | 0 minutes (immediately) post-intervention, 45 minutes post-intervention
  Rating scale, 0-100 scale with question "I think that the speaker is _____", with endpoints of "unintelligent" on the zero side and "intelligent" on the 100 side. Higher scores mean a better outcome. The Attitude Survey measures participants' knowledge, beliefs, and emotions relating to listening to a speaker with aphasia.
Rating of speaker with aphasia's language skills on the Attitude Survey | 0 minutes (immediately) post-intervention, 45 minutes post-intervention
  Rating scale, 0-100 scale with question "I think that it was _____ for the speaker to find the words for what they wanted to say", with endpoints of "hard" on the zero side and "easy" on the 100 side. Lower scores mean a better outcome. The Attitude Survey measures participants' knowledge, beliefs, and emotions relating to listening to a speaker with aphasia.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Mack, PhD, Principal Investigator — University of Massachusetts, Amherst
Locations (1):
- UMass Amherst Henry M. Thomas III Center at Springfield, Springfield, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Data to be generated from this project include language processing data collected through eye-tracking, comprehension accuracy data (mouse-click responses), and participants' responses to a survey measuring their attitudes.
  De-identified raw survey data and comprehension accuracy data will be preserved and shared. Deidentified, preprocessed eye-tracking data will be preserved and shared.
Supporting Information: Study Protocol
Time Frame: De-identified data will be available upon publication of related work or the end of the project period, whichever comes first, and will remain available indefinitely.
Access Criteria: IPD and supporting information will be freely available on Open Science Framework.